CLINICAL TRIAL: NCT01239836
Title: Self-management, Constructivism or Both as Knowledge Transfer Strategies for Reducing the Cost and Impact of Urinary Incontinence Among Community-dwelling Senior Women in the United Kingdom
Brief Title: Effectiveness of Continence Promotion Interventions Among Community-dwelling Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Brunel University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Cara Tannenbaum, Dr., Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: CIHR-200909-CUK-202417
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence, self-management, cost, self-efficacy, continence promotion
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Self-management (Experimental)
  Interventions: Behavioral: Evidence-based self-management tool
- General Health Lecture (Sham Comparator)
  Interventions: Behavioral: General health lecture
- Combined workshop and self-management (Experimental)
  Interventions: Behavioral: Constructivist interactive workshop on urinary incontinence; Behavioral: Evidence-based self-management tool
- Workshop (Experimental)
  Interventions: Behavioral: Constructivist interactive workshop on urinary incontinence

INTERVENTIONS:
Behavioral: Constructivist interactive workshop on urinary incontinence — A one hour interactive group workshop aimed at contradicting commonly held beliefs and maladaptive practices about incontinence. The interactive continence workshop was designed to create cognitive dissonance and challenge these beliefs and practices, as well as to promote more effective therapeutic strategies for correcting urine leakage.
  Arms: Combined workshop and self-management; Workshop
Behavioral: Evidence-based self-management tool — Participants will receive a customized evidence-based risk factor modification self-management tool targeting up to 6 risk factors and associated therapeutic strategies. The six risk factors are pelvic floor muscle weakness, consumption of caffeinated drinks, obesity, constipation, vision loss and smoking.
  Arms: Combined workshop and self-management; Self-management
Behavioral: General health lecture — Participants will attend a lecture on general women's health issues that does not address urinary incontinence.
  Arms: General Health Lecture

SUMMARY:
Urinary incontinence is a common and bothersome condition that remains frequently untreated among senior women. The aim of this trial is to compare the effectiveness of two community-based continence promotion interventions aimed at improving rates of self-care and/or professional health-care seeking in older women with urinary incontinence. The main hypothesis posits that participation in a constructivist interactive workshop combined with use of an evidence-based self-management tool will yield rates of improvement in incontinence frequency and reduce the cost of pad use by 20% compared to either intervention alone, which individually are expected to yield minimal effect sizes of at least 0.3 compared to a sham intervention.

DETAILED DESCRIPTION:
The research design is a 2x2 factorial open-label cluster randomised controlled trial. The cluster (unit of randomization) is at the level of each local community senior's group, from whence participants will be recruited. Incontinent community-dwelling older women aged 60 years and older who have not sought care for their urinary symptoms in the last two years, but who experience incontinence at least twice weekly will be recruited through local community organizations. Eligible participants from each local community centre will be randomly assigned as a group to one of four interventions. The first intervention is participation in an interactive constructivist continence workshop. The second intervention involves receipt of an evidence-based self-management tool for incontinence. The third group will receive both interventions. The fourth group will act as the control group: they will simply be asked about their urinary symptoms and given a general talk on women's health. At the end of the study, the control group will be offered the self-management tool.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 60 years or older
* Urinary incontinence twice weekly
* Women who have not sought medical advice for incontinence symptoms in the last 2 years.
* Fluent in English

Exclusion Criteria:

* Women who have received treatment for their urinary incontinence within the past two years from a health care provider with expertise in urinary incontinence management (i.e. nurse practitioners/physicians/surgeons who have a clinical practice that focuses on treating urinary incontinence).
* Women started on medications for urinary incontinence (i.e. antimuscarinic medication) within the 6 months prior to enrolment.
* Women with a history of a neurological condition (e.g. Multiple Sclerosis and spinal cord injury) because they require further investigation. Women identified to have these historical findings will be advised to speak to their physician immediately about their incontinence and the possible need for investigation.
* Women who do not consent to participate.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Incontinence frequency | 3 months
  Reductions in incontinence frequency as indicated on a 72-hour voiding diary at 3-months post-intervention compared to baseline.

SECONDARY OUTCOMES:
Cost of pad use | 3 months
  Reductions in the cost of pad use per day at 3-months post intervention compared to baseline.
Self-efficacy for managing incontinence | 3-months
  An increase of 5 points or more on the Geriatric Self-Efficacy index for urinary incontinence at 3-months post-intervention compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Tannenbaum, MD, Principal Investigator — Centre de recherche de l'Institut universitaire de gériatrie de Montréal; Eleanor van den Heuvel, PhD, Study Director — Brunel University
Locations (1):
- Brunel University, Uxbridge, Middlesex, United Kingdom

REFERENCES:
- [Background] Tannenbaum C, Drali R, Holroyd-Leduc J, Richard L. Lessons learned: impact of a continence promotion activity for older community-dwelling women. Neurourol Urodyn. 2010 Apr;29(4):540-4. doi: 10.1002/nau.20800. PMID 19693950
- [Derived] Tannenbaum C, Agnew R, Benedetti A, Thomas D, van den Heuvel E. Effectiveness of continence promotion for older women via community organisations: a cluster randomised trial. BMJ Open. 2013 Dec 10;3(12):e004135. doi: 10.1136/bmjopen-2013-004135. PMID 24334159